CLINICAL TRIAL: NCT00333047
Title: A Study of Letrozole in the Treatment of Metastatic Breast Cancer in Combination With Chemotherapy
Brief Title: Letrozole in Metastatic Breast Cancer in Combination With Chemotherapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345ADE07
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer; Aromatase inhibitor; Letrozole
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

INTERVENTIONS:
Drug: Letrozole

SUMMARY:
Therapeutic interventions for patients with metastatic breast cancer are aimed at prolonging survival and improving the quality of life. The objective of this trial is to assess if an initial chemotherapy followed by an endocrine therapy leads to a longer disease-free interval as compared to chemotherapy alone.

ELIGIBILITY:
Inclusion criteria

* Histologically proven metastatic breast cancer
* Measurable disease, patients with bone only disease are not eligible
* Age ≥ 65 years
* Performance status ≤ 2 (World Health Organization)
* Estimated life expectancy under therapy of at least 3 months
* Estrogen-/progesterone-receptor status positive or unknown
* Signed informed consent

Exclusion criteria

* Prior chemo- or hormone therapy for metastatic breast cancer; prior therapy with aromatase inhibitors in the adjuvant setting
* Disease-free interval after adjuvant therapy < 1 year
* Clinical signs of central nervous system metastases
* Renal, bone marrow, or liver insufficiency
* Severe coronary heart disease, cardiac insufficiency or other severe concomitant internal diseases
* Pulmonary fibrosis/alveolitis Additional protocol-defined inclusion/exclusion criteria may apply.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24
Dates: Start 2002-07

PRIMARY OUTCOMES:
Objective response rate (complete remission, partial remission,no change, progressive disease) by clinical palpation and radiologic imaging every 3 months until disease progression

SECONDARY OUTCOMES:
Time to progression and safety and toxicity during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- Kiel, Germany